CLINICAL TRIAL: NCT06460818
Title: Surgical Sample Collection- Sampling During Uterine Surgery
Status: Completed | Type: Observational
Sponsor: PinkDx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PNK001
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Women's Health

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh and frozen tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign: tissue collection from women with benign reproductive conditions
- malignant: tissue collection from women with suspected and malignant reproductive conditions

SUMMARY:
The goal of this clinical trial is to evaluate anatomical locations for sample collection for future decisions for diagnostic test development.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent form (ICF) indicating that the participant has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, investigational plan, and other procedures.
3. Females:

   1. Aged >45 for benign and pre-malignant cases
   2. Aged >18 with positive biopsies.
4. Presence of uterus.
5. Scheduled for hysterectomy.

Exclusion Criteria:

1. Investigator site staff members directly involved in the conduct of the study and their family members or participants who are Pink Dx, Inc. employees or their family members.
2. Other acute or chronic medical or psychiatric conditions that would increase the risk associated with study participation in the judgement of the investigator.
3. Women who have undergone a hysterectomy.
4. Inability or unwillingness to sign informed consent.
5. Contraindication to surgery, including pregnancy.
6. Women who have used a tampon within 7 days of surgery.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing hysterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with optimal vaginal samples obtained during the collection process | 9 months
  Number of participants with optimal vaginal samples obtained during the collection process, including preferred anatomical location and yields and quality of samples.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mariani, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No